CLINICAL TRIAL: NCT03647852
Title: Clinical Study on Strategy for Refractory Henoch-Schönlein Purpura
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Children's Hospital of Fudan University (Other)
Collaborators: Shanghai Children's Hospital (Other); Shanghai Children's Medical Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: chfuHSP 1.0
Record Dates: First submitted 2018-08-22; First posted 2018-08-27 (Actual); Last update posted 2025-02-19 (Actual); Status verified 2025-02

CONDITIONS: Henoch-Schönlein Purpura
Keywords: severe gastrointestinal involvement
MeSH Terms: conditions — IgA Vasculitis | interventions — Methylprednisolone; Immunoglobulins, Intravenous

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Methylprednisolone group (Experimental): In this group patients will be given Methylprednisolone pulse(15-30mg/kg/d) and continued with oral prednisolone (2mg/kg/d)
  Interventions: Drug: Methylprednisolone; Drug: other basic supportive treatment
- IVIG group (Active Comparator): In this group patients will be given IVIG (2g/kg) and at the same time oral prednisolone (2mg/kg/d)
  Interventions: Drug: IVIG; Drug: other basic supportive treatment

INTERVENTIONS:
Drug: Methylprednisolone — 1.methylprednisolone pulse (15-30mg/kg/d) for 3 days with continued oral prednisolone(2mg/kg/d) 2.if the patients still complain abdominal pain and feel abdominal tenderness on the third day after intervention , patients would be given IVIG(2g/kg/d)as a change
  Arms: Methylprednisolone group
Drug: IVIG — 1. IVIG 2g/kg and oral prednisolone 2mg/kg/d 2.if the patients still complain abdominal pain and feel abdominal tenderness on the third day after intervention , patients would be given methylprednisolone pulse (15-30mg/kg/d) for 3 days
  Arms: IVIG group
Drug: other basic supportive treatment — 1. Omeprazole 0.8mg/kg.d.The maximum dose is less than 40mg per day
  2. Low molecular weight heparin calcium 50IU/kg.d

SUMMARY:
IgA vasculitis is relatively common in children,especially in Asian countries. Abdominal manifestation could be severe, including bleeding, pancreatitis,appendicitis and intestinal intussusception. Delayed diagnosis could be fatal and cause severe complications.Nowadays no guidelines for those with severe abdominal manifestations in China.However, the most used treatment is steroid. For those severe forms are methylprednisolone pulse, IVIG, immunosuppressants and blood purification. Given the fact that different strategies lead to different endings which varies in cost, adverse effect and clinical outcomes in different medical centers, it is necessary to give birth to a useful and feasible strategy. This clinical trial is a muti-center, randomized,controlled prospective study.Patients with gastrointestinal disease will be recruited in three children's medical centres in Shanghai and will be randomized to two groups: MP group and IVIG group. Cost effect and clinical outcomes will be evaluated. Blood purification will be evaluated as a remedy when MP and IVIG fail to cure.

ELIGIBILITY:
Inclusion Criteria:

1. both genders
2. age between 2-16 years old
3. IgA vasculitis with gastrointestinal involvement
4. course of disease less than 2 months
5. refractory to ordinary dosage of prednisolone (less than 2mg/kg/d）

Exclusion Criteria:

1. patients with severe sepsis
2. patients with central nervous system infection,
3. patients with severe pneumonia
4. patients with chronic infection (such as EBV, CMV, Tuberculosis)
5. patients complicated by CKD who need renal replacement therapy
6. patients suffering from severe central nervous system complications as intracranial hemorrhage or neuropathy

Ages: 2 Years to 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 150 (Estimated)
Dates: Start 2019-09-01 (Actual); Primary Completion 2026-02-27 (Estimated); Study Completion 2026-10-30 (Estimated)

PRIMARY OUTCOMES:
sustained abdominal pain relief | 3 days after treatment
  no abdominal pain complaint and no abdominal tenderness

SECONDARY OUTCOMES:
sustained abdominal pain relief | 7 days after treatment
  3 days after treatment part of the patients may fail the first assigned intervention and has to accept the alternative intervention and abdominal pain complaint and abdominal tenderness will be checked at 7 days after treatment
other treatment rather than assigned intervention | 4 weeks after treatment
  other treatment such as blood purification, the second methylprednisolone pulse, and immunosuppressant will be documented if the two interventions all failed
tolarable food type | 2 weeks after treatment
  what kind of food can be tolerant ( 0 fluid, 1 semi liquid, 2 solid )
the number of days of taking fasting | At the time of discharge
  the number of days of taking fasting will be counted at the time of discharge
Drug-related side effects | 3 days after treatment
  Side effects associated with methylprednisolone and IVIG will be recorded
hypertension | 7 days after treatment
  systolic or diastolic blood pressure greater than or equal to 95% for the age, sex, and height of the patient is considered to have 1.hypertension otherwise 0. Blood pressure will be measured with mercury blood pressure monitor.
infection | 4 weeks after treatment
  different infection types should be specified
ocular hypertension | 7 days after treatment
  1.ocular hypertension 0. no ocular hypertension. Ocular hypertension will be defined as intraocular pressure of either eye is greater greater or equal to 21mmHg
steroid-related diabetes | 3 days after treatment
  1. with steroid-related diabetes 0. no steroid-related diabetes . Steroid-related diabetes will be defined as random blood sugar is greater than 11.1 mmol/l
cost of treatment | 4 weeks after treatment
  cost of treatment will be obtained from discharge fee list
The number of days in hospital | at the time of discharge
  The number of days in hospital will be counted at the time of discharge

CONTACTS AND LOCATIONS:
Overall Officials: Li Sun, MD, Principal Investigator — Children's Hospital of Fudan University; Wenyan Huang, MD, Principal Investigator — Shanghai Children's Hospital
Locations (3):
- China (3):
  - Children's Hospital of Fudan University, Shanghai
  - Children's Hospital of Shanghai, Shanghai
  - Shanghai Children's Medical Centre, Shanghai

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code